CLINICAL TRIAL: NCT04033289
Title: The Clinical Efficacy of Hip Protection Orthosis for The Protection of Hip Dislocation in Patients With Severe Cerebral Palsy, Single Blinded, Randomized-control Trial, Multicenter Clinical Trial
Brief Title: The Clinical Efficacy of Hip Protection Orthosis for the Protection of Hip Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-1906/546/002
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Device: Hip protection orthosis
- control group (No Intervention)

INTERVENTIONS:
Device: Hip protection orthosis — Experimental group would wear hip protection orthosis over 12 hours a day for 1 year.
  Arms: experimental group

SUMMARY:
Single Blinded, Randomized-control tiral, Multicenter clinical trial

ELIGIBILITY:
Inclusion Criteria:

* GMFCE level IV or V in the Cerebral palsy
* age from 1 to 10

Exclusion Criteria:

* History of hip joint surgery
* Botulinum toxin injection to hip muscle past 3 months or expected in our study duration

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Migration index | 6 months
  Hip AP radiography

SECONDARY OUTCOMES:
Cobb's angle (') | 6 months
  using radiography, expressed by degree from 0' to 180'. The closer to 0', the better the value.
Range of motion of hip joint (') | 6 months
  Using goniometer, measure the hip and knee abduction and flexion angle expressed by degree from 0' to 180'. The closer to 180', the better the value.
Visual analog scale | 6 months
  measure the pain expressed by score from 0 to 10. The closer to 10, the higher the pain.
Likert scale (score) | immediately after wearing orthosis
  measure the satisfaction about hip protection orthosis expressed by score from 0 to 5. The closer to 5, the higher the satisfaction.
Child Health Index of Life with Disabilities (CPCHILD) | 6 months
  measure the quality of life expressed by score from 0 to 100. The higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Juseok Ryu, Phd, Study Chair — professor
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim BR, Yoon JA, Han HJ, Yoon YI, Lim J, Lee S, Cho S, Shin YB, Lee HJ, Suh JH, Jang J, Beom J, Park Y, Choi JH, Ryu JS. Efficacy of a Hip Brace for Hip Displacement in Children With Cerebral Palsy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2240383. doi: 10.1001/jamanetworkopen.2022.40383. PMID 36331502